CLINICAL TRIAL: NCT05705713
Title: First-day Computed Tomography: Does it Has a Role in the Assessment of Patients With Inhalation Lung Injury?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal A. El-Koa, principle investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12/2022COM2
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Inhalation Injury
Keywords: inhalation injury; Bronchial wall thickening; Radiologist score; computed tomography.

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Experimental): 48 participants with burn injuries associated with inhalation lung injuries were recruited from the burn department.
  Interventions: Radiation: chest computed tomography (CT)
- Control (Active Comparator): 10 participants with burn injuries NOT associated with inhalation lung injuries were recruited from the burn department.
  Interventions: Radiation: chest computed tomography (CT)

INTERVENTIONS:
Radiation: chest computed tomography (CT) — Within the first 12 hours of suspected inhalation lung injury, fiberoptic bronchoscopy was done to confirm the diagnosis. After confirming the diagnosis, an initial chest CT in the first 24 hrs through which the radiologist score (RADS) together with bronchial wall thickening (BWT) was done.

SUMMARY:
A major risk factor for death in burn victims is inhalation lung injury. Diagnostic criteria and severity grading are not well understood. After an inhalation injury, the mucociliary escalator is impaired by induced mucosal hyperemia, which includes Edema, increased mucous production, and airway exudation, and these insults worsen airway narrowing which interferes with ventilation. Multimodal therapy and quick bronchoscopic diagnosis improve patient outcomes. Early identification and classification of inhalation injuries improve patient outcomes. Chest CT may be employed as an alternative to or supplement to the bronchoscopy as well as a diagnostic and prognostic tool. In this study, the diagnostic and prognostic value of bronchial wall thickening as a radiological CT finding in inhalation lung damage and the radiologist score (RADS) were evaluated.

DETAILED DESCRIPTION:
Forty-eight patients with inhalation lung injury were included in the study as the case group, and ten patients without ILI were chosen as the control group. Both groups were recruited from the burn and plastic department. A fiberoptic bronchoscope was performed during the first 12 hours of a suspected ILI to confirm the diagnosis. After performing an initial chest X-ray, computed tomography was used to calculate the radiologist score (RADS) and the thickness of the bronchial walls (BWT).

ELIGIBILITY:
Inclusion Criteria:

* any patient with a suspected inhalational lung injury

Exclusion Criteria:

* less than 18 years old,
* patients who had their CT scan after 24 hours after their admission
* patients who couldn't finish all of the study steps.
* patients that are known to have any parenchymal lung disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
bronchial wall thickening (BWT) | 24 hours
  measured through a CT chest scan at the end inspiration 2 cm distal to the tracheal bifurcation.
Radiologist score | 24 hours
  CT scans of each patient were examined using 1-cm axial slices from the apex to the diaphragm level. The right and left lung fields in each slice were subdivided into 4 quadrants. Each quadrant was awarded a score ranging from 0 to 3 based on the severity of the results. The highest score inside a quadrant was awarded as the final score, and a total score was produced for each slice. The total score for each slice was then added together for the full CT scan to get the RADS overall.

REFERENCES:
- [Background] Latenser BA, Miller SF, Bessey PQ, Browning SM, Caruso DM, Gomez M, Jeng JC, Krichbaum JA, Lentz CW, Saffle JR, Schurr MJ, Greenhalgh DG, Kagan RJ. National Burn Repository 2006: a ten-year review. J Burn Care Res. 2007 Sep-Oct;28(5):635-58. doi: 10.1097/BCR.0B013E31814B25B1. No abstract available. PMID 17969244
- [Background] Foncerrada G, Culnan DM, Capek KD, Gonzalez-Trejo S, Cambiaso-Daniel J, Woodson LC, Herndon DN, Finnerty CC, Lee JO. Inhalation Injury in the Burned Patient. Ann Plast Surg. 2018 Mar;80(3 Suppl 2):S98-S105. doi: 10.1097/SAP.0000000000001377. PMID 29461292
- [Background] Kimura R, Traber LD, Herndon DN, Linares HA, Lubbesmeyer HJ, Traber DL. Increasing duration of smoke exposure induces more severe lung injury in sheep. J Appl Physiol (1985). 1988 Mar;64(3):1107-13. doi: 10.1152/jappl.1988.64.3.1107. PMID 3366733
- [Background] Albright JM, Davis CS, Bird MD, Ramirez L, Kim H, Burnham EL, Gamelli RL, Kovacs EJ. The acute pulmonary inflammatory response to the graded severity of smoke inhalation injury. Crit Care Med. 2012 Apr;40(4):1113-21. doi: 10.1097/CCM.0b013e3182374a67. PMID 22067627
- [Background] Hassan Z, Wong JK, Bush J, Bayat A, Dunn KW. Assessing the severity of inhalation injuries in adults. Burns. 2010 Mar;36(2):212-6. doi: 10.1016/j.burns.2009.06.205. Epub 2009 Dec 16. PMID 20006445
- [Background] Oh JS, Chung KK, Allen A, Batchinsky AI, Huzar T, King BT, Wolf SE, Sjulin T, Cancio LC. Admission chest CT complements fiberoptic bronchoscopy in prediction of adverse outcomes in thermally injured patients. J Burn Care Res. 2012 Jul-Aug;33(4):532-8. doi: 10.1097/BCR.0b013e318237455f. PMID 22210063
- [Background] Walker PF, Buehner MF, Wood LA, Boyer NL, Driscoll IR, Lundy JB, Cancio LC, Chung KK. Diagnosis and management of inhalation injury: an updated review. Crit Care. 2015 Oct 28;19:351. doi: 10.1186/s13054-015-1077-4. PMID 26507130
- [Background] Yamamura H, Kaga S, Kaneda K, Mizobata Y. Chest computed tomography performed on admission helps predict the severity of smoke-inhalation injury. Crit Care. 2013 May 25;17(3):R95. doi: 10.1186/cc12740. PMID 23706091
- [Background] Charles WN, Collins D, Mandalia S, Matwala K, Dutt A, Tatlock J, Singh S. Impact of inhalation injury on outcomes in critically ill burns patients: 12-year experience at a regional burns centre. Burns. 2022 Sep;48(6):1386-1395. doi: 10.1016/j.burns.2021.11.018. Epub 2021 Nov 26. PMID 34924231
- [Background] Yamamura H, Morioka T, Hagawa N, Yamamoto T, Mizobata Y. Computed tomographic assessment of airflow obstruction in smoke inhalation injury: Relationship with the development of pneumonia and injury severity. Burns. 2015 Nov;41(7):1428-34. doi: 10.1016/j.burns.2015.06.008. Epub 2015 Jul 15. PMID 26187056
- [Background] Kim CH, Woo H, Hyun IG, Song WJ, Kim C, Choi JH, Kim DG, Lee MG, Jung KS. Pulmonary function assessment in the early phase of patients with smoke inhalation injury from fire. J Thorac Dis. 2014 Jun;6(6):617-24. doi: 10.3978/j.issn.2072-1439.2014.04.11. PMID 24976982